CLINICAL TRIAL: NCT01387113
Title: Expanding the Time Window for IV Thrombolysis With Rt-PA in Acute Ischemic Stroke Patients Using Computed Tomography Perfusion Imaging: The PERFusion Use in Stroke Evaluation (PERFUSE) Study
Brief Title: The PERFusion Use in Stroke Evaluation Study
Acronym: PERFUSE
Status: Completed | Type: Observational
Sponsor: California Pacific Medical Center Research Institute (Other)
Collaborators: California Pacific Medical Center (Other)
Responsible Party: Principal Investigator, Nobl Barazangi, Medical Doctor, California Pacific Medical Center Research Institute
Other Study IDs: PERFUSE
Record Dates: First submitted 2011-06-21; First posted 2011-07-04 (Estimated); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Ischemic Stroke
Keywords: stroke; tPA; Thrombolysis; rt-PA; Ischemic; CTP; Imaging; CT Perfusion Imaging; Perfusion; CTA; CT Angiography; Acute ischemic stroke; Acute stroke therapy; (AIS)
MeSH Terms: conditions — Ischemic Stroke; Stroke; Ischemia | interventions — Cytidine Triphosphate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute ischemic stroke patients: All acute ischemic stroke patients receiving IV rt-PA within 6 hours of symptom onset
  Interventions: Other: Computed tomography perfusion imaging

INTERVENTIONS:
Other: Computed tomography perfusion imaging — As per standard of care at CPMC

SUMMARY:
This is an open label single center phase II trial, evaluating the utility of 64 slice CT perfusion (CTP) in acute ischemic stroke (AIS) patients. The main aim is to determine which aspects of CTP imaging can aid in expanding the time window for thrombolysis with IV (rt-PA) in AIS patients up to 6 hours after symptom onset.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke
* ≥ 18 years old
* presentation up to 6 hours from time of onset of acute stroke symptoms

Exclusion Criteria:

* pregnancy
* inability to receive CT scan
* allergy to IV contrast
* symptoms with full resolution
* intracerebral hemorrhage
* severe stroke which is classified as 'malignant' (hypodensity on noncontrast CT greater than 1/3 cerebral hemisphere)
* premorbid mRS of >3
* life expectancy of ≤3 months
* any condition which, in the opinion of the investigator makes the subject unsuitable for study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All acute ischemic stroke patients who present to the emergency room at CPMC who receive IV rt-PA within 6 hours of symptom onset
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2011-05; Primary Completion 2022-07 (Actual); Study Completion 2022-07 (Actual)

PRIMARY OUTCOMES:
Final infarct volume | 24 hour post-thrombolysis

SECONDARY OUTCOMES:
Large vessel occlusion on neuroimaging | 24 hours post-thrombolysis
NIHSS | 24-hours from tPA adminsitration
Symptomatic intracerebral hemorrhage post-thrombolysis | 24 hours post-thrombolysis
Modified Rankin Scale | 3-months from tPA administration

CONTACTS AND LOCATIONS:
Overall Officials: Nobl Barazangi, MD, PhD, Principal Investigator — CPMC
Locations (1):
- California Pacific Medical Center, San Francisco, California, United States

REFERENCES:
- See also: Related Info — http://www.cpmc.org/professionals/research/trials/neurocriticalcare.html